CLINICAL TRIAL: NCT05701917
Title: DEFIANCE - ClotTriever® Thrombectomy System vs. Anticoagulation Alone for Treatment of Deep Vein Thrombosis
Brief Title: DEFIANCE: RCT of ClotTriever System Versus Anticoagulation In Deep Vein Thrombosis
Acronym: DEFIANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-001
Record Dates: First submitted 2023-01-06; First posted 2023-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Post-Thrombotic Syndrome
Keywords: Venous Thromboembolism; Deep Venous Thrombosis; Post-Thrombotic Syndrome; Anticoagulation; Percutaneous Mechanical Thrombectomy
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Postthrombotic Syndrome | interventions — Warfarin; Rivaroxaban; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Interventional (Active Comparator): Interventional strategy using the ClotTriever System to achieve and maintain vessel patency (ClotTriever Intervention Arm).
  Interventions: Device: ClotTriever System
- Conservative Medical Management (Active Comparator): Conservative medical management using anticoagulation therapy alone (Conservative Medical Management Arm).
  Interventions: Drug: Commercially available/market approved anticoagulation medication including but not limited to: Heparin Sodium, Coumadin, Rivaroxaban, Apixaban, etc.

INTERVENTIONS:
Device: ClotTriever System — Mechanical thrombectomy
  Arms: Interventional
Drug: Commercially available/market approved anticoagulation medication including but not limited to: Heparin Sodium, Coumadin, Rivaroxaban, Apixaban, etc. — Anticoagulants are a group of medications that decrease your blood's ability to clot.
  Arms: Conservative Medical Management

SUMMARY:
This study is a prospective, multicenter, randomized controlled trial of an interventional strategy using the ClotTriever System to achieve and maintain vessel patency (ClotTriever Intervention Arm) versus conservative medical management using anticoagulation therapy alone (Conservative Medical Management Arm) in the treatment of subjects with symptomatic unilateral iliofemoral DVT. The study will collect data on demographics, comorbidities, details from the DVT diagnosis and treatment, and clinical outcomes through the 6-month follow up visit.

DETAILED DESCRIPTION:
The study will compare the clinical outcomes of patients treated with an interventional strategy using the ClotTriever System to achieve and maintain vessel patency (ClotTriever Intervention Arm) versus conservative medical management using anticoagulation therapy alone (Conservative Medical Management Arm) in the treatment of symptomatic unilateral iliofemoral DVT. Approximately 300 subjects will be enrolled and randomized. All subjects who sign informed consent and who meet all of the inclusion criteria and none of the exclusion criteria will be randomized (1:1, ClotTriever Intervention Arm or Conservative Medical Management Arm).

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Proximal lower extremity unilateral DVT involving at least the common femoral, external iliac, or common iliac veins, alone or in combination
* Symptom onset within 12 weeks of enrollment in the study
* Significant symptoms, as defined by a Villalta score > 9
* Willing and able to provide informed consent

Exclusion Criteria

* Bilateral iliofemoral DVT
* Prior venous stent in the target venous segment
* IVC aplasia/hypoplasia or other congenital anatomic anomalies of the IVC or iliac veins
* IVC filter in place at the time of enrollment
* Limb-threatening circulatory compromise (e.g., phlegmasia)
* Clot in transit including IVC thrombus presenting as extension of >2cm into the IVC from the CIV
* Symptomatic PE with right heart strain where the physician judges that a DVT intervention is inappropriate at this time.
* Inability to be a candidate for intervention due to medical or technical reasons based on physician judgement
* Severe allergy, hypersensitivity to, or thrombocytopenia from heparin
* Severe allergy to iodinated contrast agents that cannot be mitigated
* Hemoglobin < 8.0 g/dL, INR > 1.7 before warfarin was started, or platelets < 50,000/µl which cannot be corrected prior to enrollment
* Severe renal impairment (estimated GFR < 30 ml/min) in patients who are not yet on dialysis
* Inability to provide therapeutic anticoagulation per Investigator discretion
* Uncontrolled severe hypertension on repeated readings (systolic > 180mmHg or diastolic > 105mmHg)
* Recently (< 30 days) had DVT interventional procedure
* Subject is participating in another study that may interfere with this study
* Life expectancy < 6 months or chronic non-ambulatory status
* Known hypercoagulable states that, in the opinion of the Investigator, cannot be medically managed throughout the study period
* Subject has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject (e.g., contraindication to use of ClotTriever per local approved labeling, compromise the well-being or that could prevent, limit, or confound the protocol-specified assessments)
* Subject has previously completed or withdrawn from this study
* Patient unwilling or unable to conduct the follow up visits per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Composite clinical endpoint constructed as a win ratio, a hierarchy of the following: | 180 Days (+-14 Days)
  1. Occurrence of treatment failure or therapy escalation
  2. Assessment of PTS severity, as defined by the Villalta scale

SECONDARY OUTCOMES:
Composite clinical endpoint constructed as a win ratio, a hierarchy of the following: | 10 Days (+- 3 Days)
  1. Vessel compressibility assessed by duplex ultrasound
  2. Pain as assessed by the NPRS
  3. An improvement of edema as assessed by leg calf circumference measurements
Assessment of PTS Severity: | 180 Days (+-14 Days)
  a. Assessment of PTS severity, as defined by the Villalta scale

CONTACTS AND LOCATIONS:
Overall Officials: Steven Abramowitz, MD, Principal Investigator — MedStar Health Research Institution; Xhorlina Marko, MD, Principal Investigator — Henry Ford Health; Stephen Black, MD, Principal Investigator — St Thomas' Hospital (UK)
Locations (63):
- United States (47):
  - Honor Health, Scottsdale, Arizona
  - Pima Heart and Vascular, Tucson, Arizona
  - UCI Medical Center, Orange, California
  - Vascular and Interventional Specialists of Orange County, Orange, California
  - University Of Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Health Research Institution, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Lakeland Vascular Institute, Lakeland, Florida
  - HCA Florida Largo Hospital, Largo, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - BayCare Health System, Tampa, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Community Healthcare System, Munster, Indiana
  - St. Elizabeth Edgewood, Edgewood, Kentucky
  - University of Maryland, Baltimore, Maryland
  - McLaren Healthcare, Bay City, Michigan
  - Henry Ford Health, Detroit, Michigan
  - MyMichigan Medical Center, Midland, Michigan
  - University of Missouri, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Northwell Health, Bay Shore, New York
  - NYP-Brooklyn Methodist, Brooklyn, New York
  - SUNY, The University at Buffalo, Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Mission Health, Asheville, North Carolina
  - Mercy Health - The Heart Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Saint Francis Hospital, Tulsa, Oklahoma
  - Allegheny St. Vincent Hospital, Erie, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Health Research Network, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Upstate, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Clements University Hospital (UTSW), Dallas, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Providence Sacred Heart Med Center, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Vienna General Hospital (AKH Wien), Vienna, Austria
- Helsinki University Hospital, Helsinki, Finland
- Germany (7):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Würtemberg
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt am Main, Hesse
  - Klinikum Hochsauerland GmbH, Arnsberg, North Rhine-Westphalia
  - Universität Leipzig, Leipzig, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Heidelberg, Heidelberg
- Switzerland (3):
  - Kantonsspital Baden, Baden
  - Inselspital, Universitätsspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne
- United Kingdom (4):
  - GSST London/St Thomas, London
  - Imperial College, London
  - Freeman Hospital Newcastle upon Tyne, Newcastle upon Tyne
  - Oxford - John Radcliffe, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abramowitz SD, Marko X, D'Souza D, Noor S, Pereira K, Silver MJ, Rosenberg SP, Markovitz CD, Tu T, Weinberg I, Black S. Rationale and design of the DEFIANCE study: A randomized controlled trial of mechanical thrombectomy versus anticoagulation alone for iliofemoral deep vein thrombosis. Am Heart J. 2025 Mar;281:92-102. doi: 10.1016/j.ahj.2024.10.016. Epub 2024 Nov 3. PMID 39491572
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829